CLINICAL TRIAL: NCT06987669
Title: Gastric Emptying Assessed by Gastric Ultrasound (US) in Healthy Volunteers and Semaglutide Users: Cohort Study
Brief Title: Gastric Emptying in Healthy Volunteers and GLP-1 Agonist Users
Acronym: aGLP1-GUS
Status: Not yet recruiting | Type: Observational
Sponsor: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, Javiera Vargas, Medical Doctor, Clinica Alemana de Santiago
Other Study IDs: ID1406; 2024-100 (Other: Comité Etico Cientifico Facultad de Medicina Universidad del Desarrollo Clínica Alemana)
Record Dates: First submitted 2025-05-08; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Type 2; Obesity and Overweight
Keywords: agonist GLP-1; perioperative fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers after high fat standardized breakfast: GUS will be made
  Interventions: Diagnostic Test: Gastric Ultrasound
- Patients on GLP-1 agonist: Patients on GLP-1 agonist after clear fluids diet of 18/24 hrs. GUS will be made.
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — A gastric ultrasound will be performed to determine the state of the stomach. Empty, clear fluids, solid, and in case of fluid, the amount of it ( using free tracing)
  Other Names: GUS

SUMMARY:
This observational study aims to determine the gastric emptying kinetics assessed by ultrasound in healthy volunteers after a standard breakfast and the state of the stomach after a clear liquid diet for 18 /24 hours in patients on GLP-1 agonist. The main questions it seeks to answer are:

* Is the kinetic after a standard breakfast that includes ( avocado and eggs: high fat) as fast as a standard meal that does not involve this food?
* Is a clear liquid diet of 18 to 24 hours enough to be an empty-stomach, assessed by Ultrasound in patients on GLP1 agonist?

Participants will be asked to do:

-A baseline Gastric US will be performed for healthy volunteers, and then they will have a standardized breakfast. An hourly or bihourly assessment will be done by the US.

DETAILED DESCRIPTION:
GLP-1 analogues enhance insulin secretion from β-cells, reduce glucagon secretion, have an appetite-suppressing effect, and delay gastric emptying. This last effect may make standard preoperative fasting inadequate, compromising airway safety during elective surgery and increasing aspiration risk.

The main goal is to gather evidence to determine the optimal fasting period and dietary regimen to ensure safe outpatient surgery without increasing the risk of aspiration.Ultrasound gastric content assessment is a highly accessible, bedside, cost-free, and low-risk tool for anesthesiologists. The increased use of these drugs in surgical patients and the lack of international consensus on their discontinuation and fasting protocols before surgery necessitate further study. Our hypothesis is that GLP-1 analogue users (for weight loss or diabetes) have significantly slower gastric emptying, but a 24-hour liquid regimen may be sufficient to ensure an empty stomach and safe elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Healthy volunteers or semaglutide users

Exclusion Criteria:

* Bariatric surgery
* Hiatal hernia
* Impairment to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be assessed for emptying the stomach after a standardized high-fat meal, by ultrasound.
  Cohort of patients on a GLP-1 agonist after 18/24 hours of clear fluids.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2025-05-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with each Grade ( stomach content characteristics) according Perlas et al | 24 hours tops since the starting of the clear fluid diet
  Grade 0 ( empty in supine and RLD), Grade 1 ( empty supine but liquid content on RDL), Grade 3 ( Solid content or fluid with an area of more than or equal to 10 cm2).

SECONDARY OUTCOMES:
Area of the stomach in supine and in RLD assessed by ultrasound | 24 hours tops since the starting of the clear fluid diet
  Grade 0 ( empty in supine and RLD), Grade 1 ( empty supine but liquid content on RDL), Grade 3 ( Solid content or fluid with an area of more than or equal to 10 cm2).

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, MSc, Study Chair — Universidad de Toronto; Juan Pablo Ghiringelli, Study Director — Universidad de Valparaiso; Miguel vega, MD, Study Director — Universidad del Desarrollo